CLINICAL TRIAL: NCT03195335
Title: Validity and Reliability of Turkish Version of LIFE Habits (Life-H) Assessment for Children With Cerebral Palsy
Brief Title: Turkish Version of LIFE Habits Assessment
Acronym: TVoLHA
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Collaborators: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Mintaze Kerem Gunel, Prof. Doc. Dr., Hacettepe University
Other Study IDs: 116S359
Record Dates: First submitted 2017-06-16; First posted 2017-06-22 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Participation; LIFE Habits (life-H); Validity; Reliability
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with cerebral palsy: Children who diagnosed as cerebral palsy by a pediatric neurologist
  Interventions: Other: Assessment via questionnaire

INTERVENTIONS:
Other: Assessment via questionnaire — All the children will be assessed via assessment questionnaires.

SUMMARY:
Cerebral Palsy (CP) is the most common cause of physical disability in children, is a non-progressive neurological impairment resulting from an injury in the developing brain and causing various problems related to sensory, perception, cognition, and movement. This problems leads activity and participation levels of the children with CP. In the literature various assessment tools developed for assessing participation. Assessment of Life Habits (LIFE-H) questionnaire is one of the assessment tools that examines activities of daily life and participation in detail. The scale is originally in French but English and German versions are also available. The aim of this study is to translate the scale to Turkish and to determine validity and reliability of Turkish version of Life Habits questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* To be diagnosed as cerebral palsy

Exclusion Criteria:

* Children whose family didn't accept to participate to study

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The subjects will be recruited from children who lives in Ankara city and, attend special education centers.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Life Habits Questionnaire (LIFE-H) | At baseline
  Assessing of the participation level of children

SECONDARY OUTCOMES:
Gross Motor Function Classification System (GMFCS) | At baseline
  Assessing severity of the disability of children
Pediatric Outcomes Date Collection (PODCI) (Questionnaire) | At baseline
  Assessing health-related quality of life of children by parent proxy questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Mintaze KEREM GÜNEL, Principal Investigator — Prof. Dr.
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Noreau, Luc, Patrick Fougeyrollas, and Claude Vincent.
- [Background] Damiano, Diane L., Marc D. Gilgannon, and Mark F. Abel.